CLINICAL TRIAL: NCT04032093
Title: A PHASE 2B, RANDOMIZED, PLACEBO-CONTROLLED, OBSERVER-BLINDED TRIAL TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A RESPIRATORY SYNCYTIAL VIRUS (RSV) VACCINE IN PREGNANT WOMEN 18 THROUGH 49 YEARS OF AGE AND THEIR INFANTS
Brief Title: A PHASE 2B PLACEBO-CONTROLLED, RANDOMIZED STUDY OF A RESPIRATORY SYNCYTIAL VIRUS (RSV) VACCINE IN PREGNANT WOMEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C3671003
Record Dates: First submitted 2019-07-22; First posted 2019-07-25 (Actual); Results first posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Respiratory Tract Infection
Keywords: Respiratory tract infection; Respiratory Syncytial Virus; RSV; Vaccine
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Respiratory Syncytial Virus Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is an observer-blinded study. Study staff dispensing and administering the vaccine will be unblinded, but the participant and all other study personnel, including the principal investigator, will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- RSV dose with aluminum hydroxide (Experimental): RSV vaccine with aluminum hydroxide
  Interventions: Biological: RSV vaccine
- RSV dose without aluminum hydroxide (Experimental): RSV vaccine without aluminum hydroxide
  Interventions: Biological: RSV vaccine
- Higher RSV dose with aluminum hydroxide (Experimental): Higher dose level RSV vaccine with aluminum hydroxide
  Interventions: Biological: RSV vaccine
- Higher RSV dose without aluminum hydroxide (Experimental): Higher dose level RSV vaccine without aluminum hydroxide
  Interventions: Biological: RSV vaccine
- Placebo dose (Placebo Comparator): Normal saline solution for injection (0.9% sodium chloride injection)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSV vaccine — RSV vaccine
  Arms: Higher RSV dose with aluminum hydroxide; Higher RSV dose without aluminum hydroxide; RSV dose with aluminum hydroxide; RSV dose without aluminum hydroxide
Biological: Placebo — Normal saline solution for injection (0.9% sodium chloride injection)
  Arms: Placebo dose

SUMMARY:
This Phase 2b study will evaluate the safety, tolerability, and immunogenicity of an RSV vaccine in pregnant participants who receive either one of 2 dose levels of the vaccine, formulated with or without aluminum hydroxide, or placebo, and investigate safety and characteristics of antibodies in their infants.

DETAILED DESCRIPTION:
This Phase 2b, multicenter, randomized, placebo-controlled study will evaluate the safety, tolerability, and immunogenicity of a respiratory syncytial virus stabilized prefusion F subunit vaccine (RSV vaccine) in pregnant participants who receive either one of 2 dose levels of the vaccine, formulated with or without aluminum hydroxide, or placebo, as well as assess safety and characteristics of transplacentally transferred antibodies in their infants.

ELIGIBILITY:
Inclusion Criteria - Maternal participants:

* Healthy women 18 to 49 years of age between 24 and 36 weeks of gestation on the day of planned vaccination, with an uncomplicated pregnancy, who are at no known increased risk for complications, and whose fetus has no significant abnormalities observed on ultrasound.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Receiving prenatal standard of care.
* Had an ultrasound performed at >=18 weeks of pregnancy.
* Had a negative urinalysis for protein and glucose at the screening visit. Trace protein in the urine is acceptable if the blood pressure is also normal.
* Determined by medical history, physical examination, screening laboratory assessment, and clinical judgment to be appropriate for inclusion in the study.
* Documented negative human immunodeficiency virus antibody, hepatitis B virus surface antigen, hepatitis C virus antibody, and syphilis tests at the screening visit.
* Body mass index of </=40 kg/m2 at the time of the screening visit.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent document and in this protocol.
* Expected to be available for the duration of the study and willing to give informed consent for her infant to participate in the study.

Inclusion Criteria - Infant Participants:

* Evidence of a signed and dated ICD signed by the parent(s).
* Parent(s) willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria - Maternal Participants:

* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction to any component of the investigational product or any related vaccine.
* History of latex allergy.
* History of any severe allergic reaction.
* Participants with known or suspected immunodeficiency.
* Current pregnancy resulting from in vitro fertilization or other assisted reproductive technology.
* A prior history of or known current pregnancy complications or abnormalities that will increase the risk associated with the participant's participation in and completion of the study.
* Major illness of the mother or conditions of the fetus that, in the investigator's judgment, will substantially increase the risk associated with the participant's participation in, and completion of, the study or could preclude the evaluation of the participant's response.
* Participant with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention including but not limited to systemic or cutaneous lupus erythematosus, autoimmune arthritis/rheumatoid arthritis, Guillain-Barré syndrome, multiple sclerosis, Sjögren's syndrome, idiopathic thrombocytopenia purpura, glomerulonephritis, autoimmune thyroiditis, giant cell arteritis (temporal arteritis), psoriasis, and insulin-dependent diabetes mellitus (type 1).
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Participation in other studies involving investigational drug(s) within 28 days prior to study entry and/or during study participation.
* Participants who receive treatment with immunosuppressive therapy including cytotoxic agents or systemic corticosteroids (such as for cancer or an autoimmune disease), or planned receipt of such treatment or agents during study participation. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, participants should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 30 days before investigational product administration. Inhaled/nebulized, intra articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
* Current alcohol abuse or illicit drug use.
* Receipt of blood or plasma products or immunoglobulin, from 60 days before investigational product administration, or planned receipt through delivery, with 1 exception, Rho(D) immune globulin (eg, RhoGAM), which can be given at any time.
* Previous vaccination with any licensed or investigational RSV vaccine or planned receipt during study participation.
* Laboratory test results at the screening visit outside the normal reference value for pregnant women according to their trimester in pregnancy.
* Participants who are breastfeeding at the time of the screening visit.

Exclusion Criteria - Infant Participants:

• Infant who is a direct descendant (eg, child or grandchild) of the study personnel.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy women 18 to 49 years of age who are between 24 and 36 weeks of gestation on the day of planned vaccination, with an uncomplicated pregnancy, who are at no known increased risk for complications, and whose fetus has no significant abnormalities observed on ultrasound
Enrollment: 1153 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (157):
- United States (143):
  - Children's of Alabama, Birmingham, Alabama
  - UAB Women & Infants Center - UAB Medicine, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cullman Clinical Research, Inc, Cullman, Alabama
  - Cullman Primary Care, PC, Cullman, Alabama
  - Cullman Regional, Cullman, Alabama
  - Arrowhead Hospital, Glendale, Arizona
  - Abrazo West Campus Hospital, Goodyear, Arizona
  - St. Joseph Hospital, Phoenix, Arizona
  - MedPharmics, LLC, Phoenix, Arizona
  - Mesquite Pediatrics, Tucson, Arizona
  - Watching Over Mothers and Babies, Tucson, Arizona
  - Join Clinical Trials, Bellflower, California
  - Chowchilla Hospital Clinic, Chowchilla, California
  - Join Clinical Trials, Huntington Park, California
  - Matrix Clinical Research, Huntington Park, California
  - Join Clinical Trials, Los Angeles, California
  - East Los Angeles Doctors Hospital, Los Angeles, California
  - White Memorial Medical Center, Los Angeles, California
  - Matrix Clinical Research, Los Angeles, California
  - Affiliated Physician Practice, Madera, California
  - Charles E. Ugwu-Oju, MD, FACOG, Madera, California
  - Madera Community Hospital, Madera, California
  - Madera Family Medical Group, Madera, California
  - Monterey Park Hospital, Monterey Park, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Anschutz Inpatient Pavilion 2, Aurora, Colorado
  - University of Colorado AO1, Aurora, Colorado
  - University of Colorado Hospital Inpatient Pavilion, Aurora, Colorado
  - University of Colorado Hospital Outpatient Pavilion, Aurora, Colorado
  - University of Colorado Leprino Building, Aurora, Colorado
  - University of Colorado Research II Building, Aurora, Colorado
  - Emory Children's Center, Atlanta, Georgia
  - Bingham Memorial Hospital, Blackfoot, Idaho
  - Elite Clinical Trials LLLP, Blackfoot, Idaho
  - Grove Creek Medical Center, Blackfoot, Idaho
  - Clinical Research Prime, Idaho Falls, Idaho
  - Eastern Idaho Regional Medical Center, Idaho Falls, Idaho
  - Family First Medical Center, Idaho Falls, Idaho
  - Mountain View Hospital, Idaho Falls, Idaho
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - The Pediatric Center, Idaho Falls, Idaho
  - Saltzer Medical Group, Nampa, Idaho
  - ASR, LLC, Nampa, Idaho
  - Pocatello Women's Health Clinic, Pocatello, Idaho
  - Portneuf Medical Center, Pocatello, Idaho
  - The Pediatric Center, Rigby, Idaho
  - The Iowa Clinic, Ankeny, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - The Iowa Clinic, West Des Moines, Iowa
  - Alliance for Multispecialty Research, LLC, El Dorado, Kansas
  - Hutchinson Clinic, P.A., Hutchinson, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - Cambridge Medical Trials, Alexandria, Louisiana
  - MedPharmics, LLC, Metairie, Louisiana
  - Allina Health Blaine Clinic, Blaine, Minnesota
  - Allina Health Coon Rapids Clinic, Coon Rapids, Minnesota
  - Allina Health Mercy Women's Clinic, Coon Rapids, Minnesota
  - Mercy Hospital (Allina Health), Coon Rapids, Minnesota
  - The Mother Baby Center at Mercy with Children's (Allina Health), Coon Rapids, Minnesota
  - Allina Health Fridley Clinic, Fridley, Minnesota
  - Infectious Disease Research, Minneapolis, Minnesota
  - Abbott Northwestern Hospital (Allina Health), Minneapolis, Minnesota
  - Oshsner Medical Center - Hancock, Bay Saint Louis, Mississippi
  - Merit Health Biloxi, Biloxi, Mississippi
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Gulfport OB-GYN, Gulfport, Mississippi
  - MedPharmics, LLC, Gulfport, Mississippi
  - Singing River Health System, Gulfport, Mississippi
  - St Lukes Hospital, Chesterfield, Missouri
  - Baer Pediatrics, St Louis, Missouri
  - KDB Enterprises, St Louis, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Boeson Research, Great Falls, Montana
  - Boeson Research, Missoula, Montana
  - Bryan Health, Lincoln, Nebraska
  - Bryan Women's Care Physicians, Lincoln, Nebraska
  - Midwest Childrens Health Research Institute, Lincoln, Nebraska
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - MedPharmics, Albuquerque, New Mexico
  - Winthrop Women's Wellness, Hempstead, New York
  - Sante Comprehensive Women's Healthcare, Johnson City, New York
  - NYU Winthrop Hospital, Research Pharmacy, Mineola, New York
  - NYU Winthrop Hospital, Mineola, New York
  - NYU Winthrop Pediatric Infectious Diseases, Mineola, New York
  - Women's Contemporary Care Associates, Mineola, New York
  - University of Rochester Obstetrics and Gynecology, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - Duke Children's Primary Care - Roxboro Street, Durham, North Carolina
  - Duke Regional Hospital, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Sugarcamp Family Practice, Dayton, Ohio
  - Needmore Medical Center, Dayton, Ohio
  - Kettering Medical Center, Dayton, Ohio
  - HWC Women's Center Research, Englewood, Ohio
  - Lowcountry Womens Specialists, Summerville, South Carolina
  - Summerville Medical Center, Summerville, South Carolina
  - Coastal Pediatric Research, Summerville, South Carolina
  - Center for Women''s Health and Birthcare, Beaumont, Texas
  - CHRISTUS St. Elizabeth Hospital, Beaumont, Texas
  - Gadolin Research, LLC, Beaumont, Texas
  - Pediatric Clinic of Dr. Alvin H. Prause, Beaumont, Texas
  - Texas Health Harris Methodist Hurst-Euless-Bedford Hospital, Bedford, Texas
  - Texas Health Huguley Hospital South, Burleson, Texas
  - 8th Avenue Obstetrics and Gynecology, Fort Worth, Texas
  - Baylor Scott & White of Fort Worth, Fort Worth, Texas
  - Texas Health Harris Methodist Hospital FTW, Fort Worth, Texas
  - Ventavia Research Group, LLC, Fort Worth, Texas
  - Texas Health Harris Methodist Hospital Southwest, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Chisholm Trail Pediatrics, Georgetown, Texas
  - FMC Science, LLC, Georgetown, Texas
  - Georgetown OBGYN, Georgetown, Texas
  - St. David's Georgetown Hospital, Georgetown, Texas
  - Baylor Scott & White of Grapevine (Hospital), Grapevine, Texas
  - Dr Van Tran Family Practice, Houston, Texas
  - HG Pediatrics, Houston, Texas
  - Memorial Herman Greater Heights Hospital, Houston, Texas
  - Ventavia Research Group, LLC, Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - AdventHealth Family Medicine Rural Health Clinic, Inc., Lampasas, Texas
  - FMC Science, Lampasas, Texas
  - DCOL Center For Clinical Research, Longview, Texas
  - Diagnostic Clinic of Longview, Longview, Texas
  - Longview Regional Medical Center, Longview, Texas
  - Dr. Ruben Aleman and Associates, McAllen, Texas
  - Exygon Clinical Research, Pharr, Texas
  - Texas Health Presbyterian Hospital, Plano, Texas
  - Ventavia Research Group LLC, Plano, Texas
  - Ascension Seton Williamson, Round Rock, Texas
  - Intermountain Medical Center, Murray, Utah
  - JBR Clinical Research, Salt Lake City, Utah
  - Old Farm Obstetrics & Gynecology, LLC, Salt Lake City, Utah
  - St. Marks Hospital, Salt Lake City, Utah
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Johnston Willis Hospital, Richmond, Virginia
  - Cabell Huntington Hospital, Huntington, West Virginia
  - Marshall Health dba University Pediatrics, Huntington, West Virginia
  - Marshall Health Department of Obstetrics and Gynecology, Huntington, West Virginia
  - Translational Genomic Research Institute, Huntington, West Virginia
- Argentina (2):
  - Clinica Mayo De U.M.C.B. S.R.L., San Miguel de Tucumán, Tucumán Province
  - Instituto de Maternidad y Ginecologia, Nuestra Senora de Las Mercedes, San Miguel de Tucumán, Tucumán Province
- Chile (9):
  - Hospital Base San Jose de Osorno, Osorno, Los Lagos Region
  - Hospital San Borja Arriaran, Santiago, RM
  - Clinica Universidad de los Andes, Santiago, Santiago Metropolitan
  - Instituto de Investigaciones Materno Infantil (IDIMI), Santiago, Santiago Metropolitan
  - Hospital San Jose, Santiago, Santiago Metropolitan
  - Grupo Estudios Clinicos Infectologia Respiratoria, Facultad de Medicina Universidad de Chile, Santiago, Santiago Metropolitan
  - Hospital Clinico Universidad de Chile, Santiago, Santiago Metropolitan
  - Centro Internacional de Estudios Clinicos - CIEC, Santiago, Santiago Metropolitan
  - Hospital Padre Hurtado, Santiago, Santiago Metropolitan
- New Zealand (2):
  - Christchurch Clinical Studies Trust Ltd, Christchurch
  - Christchurch Hospital (Canterbury District Health Board), Christchurch
- Respiratory and Meningeal Pathogens Research Unit (RMPRU), Soweto, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Simoes EAF, Center KJ, Tita ATN, Swanson KA, Radley D, Houghton J, McGrory SB, Gomme E, Anderson M, Roberts JP, Scott DA, Jansen KU, Gruber WC, Dormitzer PR, Gurtman AC. Prefusion F Protein-Based Respiratory Syncytial Virus Immunization in Pregnancy. N Engl J Med. 2022 Apr 28;386(17):1615-1626. doi: 10.1056/NEJMoa2106062. PMID 35476650
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671003

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pregnant maternal participants between 18 to 49 years of age and infants who were born to these maternal participants were enrolled in this study.
Pre-assignment Details: 778 maternal participants signed the informed consent form (ICF). 197 participants were screen failures who did not meet criteria and were not enrolled. 581 maternal participants and 572 infants born to maternal participants were randomized into the study.
Groups:
- Maternal Participants: RSVpreF 120 mcg: Maternal participants received a single dose of 0.5 milliliter (mL) as intramuscular injection of Respiratory Syncytial Virus prefusion F (RSVpreF) vaccine 120 mcg reconstituted with sterile water for injection on Day 1. Participants were followed up to 12 months after delivery.
- Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide: Maternal participants received a single dose of 0.5 mL as intramuscular injection of RSVpreF vaccine 120 mcg reconstituted with sterile suspension of aluminum hydroxide in water for injection on Day 1. Participants were followed up to 12 months after delivery.
- Maternal Participants: RSVpreF 240 mcg: Maternal participants received a single dose of 0.5 mL as intramuscular injection of RSVpreF vaccine 240 mcg reconstituted with sterile water for injection on Day 1. Participants were followed up to 12 months after delivery.
- Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide: Maternal participants received a single dose of 0.5 mL as intramuscular injection of RSVpreF vaccine 240 mcg reconstituted with sterile suspension of aluminum hydroxide in water for injection on Day 1. Participants were followed up to 12 months after delivery.
- Maternal Participants: Placebo: Maternal participants received a single dose of 0.5 mL as intramuscular injection of placebo (normal sterile saline solution) on Day 1. Participants were followed up to 12 months after delivery.
- Infant Participants: RSVpreF 120 mcg: Infant participants who were born to maternal participants vaccinated with RSVpreF 120 mcg (reconstituted with sterile water for injection) during pregnancy were included. Infant participants were followed up to 12 months after birth.
- Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide: Infant participants who were born to maternal participants vaccinated with RSVpreF 120 mcg (reconstituted with sterile suspension of aluminum hydroxide in water for injection) during pregnancy were included. Infant participants were followed up to 12 months after birth.
- Infant Participants: RSVpreF 240 mcg: Infant participants who were born to maternal participants vaccinated with RSVpreF 240 mcg (reconstituted with sterile water for injection) during pregnancy were included. Infant participants were followed up to 12 months after birth.
- Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide: Infant participants who were born to maternal participants vaccinated with RSVpreF 240 mcg (reconstituted with sterile suspension of aluminum hydroxide in water for injection) during pregnancy were included. Infant participants were followed up to 12 months after birth.
- Infant Participants: Placebo: Infant participants who were born to maternal participants administered with placebo (normal sterile saline solution) during pregnancy were included. Infant participants were followed up to 12 months after birth.
Period: Overall Study
Arm/Group | Maternal Participants: RSVpreF 120 mcg | Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide | Maternal Participants: RSVpreF 240 mcg | Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide | Maternal Participants: Placebo | Infant Participants: RSVpreF 120 mcg | Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide | Infant Participants: RSVpreF 240 mcg | Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide | Infant Participants: Placebo
Started | 116 | 117 | 116 | 115 | 117 | 114 | 117 | 113 | 112 | 116
Safety Set | 115 (1 maternal participant randomized to this arm but not vaccinated. Hence excluded from safety set.) | 117 | 116 | 114 (1 maternal participant randomized to this arm but not vaccinated. Hence excluded from safety set.) | 117 | 114 | 117 | 113 | 112 | 116
Completed | 107 | 107 | 108 | 100 | 99 | 106 | 107 | 108 | 100 | 98
Not Completed | 9 | 10 | 8 | 15 | 18 | 8 | 10 | 5 | 12 | 18
Not completed — Lost to Follow-up | 7 | 7 | 6 | 10 | 13 | 7 | 7 | 5 | 9 | 12
Not completed — No Longer Meets Eligibility Criteria | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 1
Not completed — Other | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Maternal safety population included all randomized maternal participants who received investigational product and were analyzed according to the investigational product they received. Infant safety population included all infant participants who were born to vaccinated maternal participants and were analyzed according to the investigational product their mothers received.
Groups:
- Maternal Participants: RSVpreF 120 mcg: Maternal participants received a single dose of 0.5 mL as intramuscular injection of RSVpreF vaccine 120 mcg reconstituted with sterile water for injection on Day 1. Participants were followed up to 12 months after delivery.
- Total: Total of all reporting groups
Arm/Group | Maternal Participants: RSVpreF 120 mcg | Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide | Maternal Participants: RSVpreF 240 mcg | Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide | Maternal Participants: Placebo | Infant Participants: RSVpreF 120 mcg | Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide | Infant Participants: RSVpreF 240 mcg | Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide | Infant Participants: Placebo | Total
Number analyzed (Participants) | 115 | 117 | 116 | 114 | 117 | 114 | 117 | 113 | 112 | 116 | 1151
Age, Customized [Count of Participants; unit: Participants]
  Less than or equal to(<=) 18 years | 0 | 0 | 0 | 0 | 0 | 114 | 117 | 113 | 112 | 116 | 572
  Greater than or equal to (>=)18 and <= 49 years | 115 | 117 | 116 | 114 | 117 | 0 | 0 | 0 | 0 | 0 | 579
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 117 | 116 | 114 | 117 | 62 | 58 | 58 | 55 | 53 | 865
  Male | 0 | 0 | 0 | 0 | 0 | 52 | 59 | 55 | 57 | 63 | 286
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 34 | 28 | 33 | 33 | 33 | 37 | 28 | 32 | 33 | 323
  Not Hispanic or Latino | 83 | 83 | 87 | 81 | 84 | 81 | 79 | 84 | 79 | 81 | 822
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 4
  Asian | 1 | 2 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 4
  Black or African American | 25 | 25 | 26 | 24 | 19 | 25 | 24 | 27 | 23 | 19 | 237
  White | 85 | 86 | 88 | 86 | 94 | 79 | 86 | 82 | 84 | 89 | 859
  More than one race | 0 | 0 | 0 | 0 | 2 | 6 | 1 | 1 | 2 | 2 | 14
  Unknown or Not Reported | 4 | 3 | 1 | 1 | 0 | 3 | 4 | 2 | 2 | 5 | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Maternal Participants With Prespecified Local Reactions by Maximum Severity Within 7 Days After Vaccination
Description: Local reactions included pain at injection site, redness and swelling and were recorded by participants in an electronic diary (e-diary). Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 centimeter (cm) and graded as mild: greater than (>) 2.0 to 5.0 cm, moderate: >5.0 to 10.0 cm and severe: >10.0 cm. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity and severe: prevented daily activity. The maximum severity was defined as highest grading of each local reaction within 7 days of vaccination.
Time Frame: Within 7 days after vaccination
Population: Maternal safety population included all randomized maternal participants who received investigational product and were analyzed according to the investigational product they received. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Maternal Participants: RSVpreF 120 mcg | Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide | Maternal Participants: RSVpreF 240 mcg | Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide | Maternal Participants: Placebo
Number analyzed (Participants) | 114 | 115 | 116 | 114 | 117
Percentage of participants
  Redness: Mild | 3.5 [1.0 to 8.7] | 2.6 [0.5 to 7.4] | 5.2 [1.9 to 10.9] | 0.9 [0.0 to 4.8] | 0 [0.0 to 3.1]
  Redness: Moderate | 0.9 [0.0 to 4.8] | 1.7 [0.2 to 6.1] | 0.9 [0.0 to 4.7] | 2.6 [0.5 to 7.5] | 0.9 [0.0 to 4.7]
  Redness: Severe | 0 [0.0 to 3.2] | 0 [0.0 to 3.2] | 0 [0.0 to 3.1] | 0 [0.0 to 3.2] | 0 [0.0 to 3.1]
  Swelling: Mild | 3.5 [1.0 to 8.7] | 2.6 [0.5 to 7.4] | 4.3 [1.4 to 9.8] | 3.5 [1.0 to 8.7] | 0.0 [0.0 to 3.1]
  Swelling: Moderate | 0.0 [0.0 to 3.2] | 2.6 [0.5 to 7.4] | 0.9 [0.0 to 4.7] | 0.9 [0.0 to 4.8] | 0.0 [0.0 to 3.1]
  Swelling: Severe | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1]
  Pain at injection site: Mild | 22.8 [15.5 to 31.6] | 53.0 [43.5 to 62.4] | 28.4 [20.5 to 37.6] | 47.4 [37.9 to 56.9] | 12.8 [7.4 to 20.3]
  Pain at injection site: Moderate | 6.1 [2.5 to 12.2] | 15.7 [9.5 to 23.6] | 5.2 [1.9 to 10.9] | 13.2 [7.6 to 20.8] | 0.0 [0.0 to 3.1]
  Pain at injection site: Severe | 0.0 [0.0 to 3.2] | 1.7 [0.2 to 6.1] | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1]

2. Primary Outcome: Percentage of Maternal Participants With Prespecified Systemic Events by Maximum Severity Within 7 Days After Vaccination
Description: Systemic events included fever, fatigue, headache, nausea, muscle pain, joint pain, vomiting, diarrhea and were recorded by participants in an e-diary. Fever was categorized as: grade 1: mild (>=38.0 to 38.4 degrees [deg] Celsius [C]), grade 2: moderate (>38.4 to 38.9 deg C), grade 3: severe (>38.9 to 40.0 deg C) and grade 4 (>40.0 deg C). Fatigue, headache, nausea, muscle pain and joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity. Vomiting was graded as mild: 1 to 2 times in 24 hours(h), moderate: >2 times in 24h and severe: required intravenous hydration. Diarrhea was graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h and severe: 6 or more loose stools in 24h. The maximum severity was defined as highest grading of each systemic event within 7 days of vaccination.
Time Frame: Within 7 days after vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Maternal Participants: RSVpreF 120 mcg | Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide | Maternal Participants: RSVpreF 240 mcg | Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide | Maternal Participants: Placebo
Number analyzed (Participants) | 114 | 115 | 116 | 114 | 117
Percentage of participants
  Fever: Grade 1 | 2.6 [0.5 to 7.5] | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1]
  Fever: Grade 2 | 0.9 [0.0 to 4.8] | 2.6 [0.5 to 7.4] | 1.7 [0.2 to 6.1] | 0.9 [0.0 to 4.8] | 0.9 [0.0 to 4.7]
  Fever: Grade 3 | 0.0 [0.0 to 3.2] | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1]
  Fever: Grade 4 | 0.0 [0.0 to 3.2] | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1]
  Fatigue: Mild | 22.8 [15.5 to 31.6] | 27.0 [19.1 to 36.0] | 23.3 [15.9 to 32.0] | 25.4 [17.7 to 34.4] | 24.8 [17.3 to 33.6]
  Fatigue: Moderate | 24.6 [17.0 to 33.5] | 17.4 [11.0 to 25.6] | 19.8 [13.0 to 28.3] | 23.7 [16.2 to 32.6] | 20.5 [13.6 to 29.0]
  Fatigue: Severe | 0.9 [0.0 to 4.8] | 3.5 [1.0 to 8.7] | 2.6 [0.5 to 7.4] | 1.8 [0.2 to 6.2] | 1.7 [0.2 to 6.0]
  Headache: Mild | 18.4 [11.8 to 26.8] | 19.1 [12.4 to 27.5] | 25.0 [17.4 to 33.9] | 18.4 [11.8 to 26.8] | 14.5 [8.7 to 22.2]
  Headache: Moderate | 10.5 [5.6 to 17.7] | 16.5 [10.3 to 24.6] | 12.1 [6.8 to 19.4] | 10.5 [5.6 to 17.7] | 9.4 [4.8 to 16.2]
  Headache: Severe | 0.0 [0.0 to 3.2] | 1.7 [0.2 to 6.1] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 1.7 [0.2 to 6.0]
  Nausea: Mild | 14.9 [8.9 to 22.8] | 17.4 [11.0 to 25.6] | 16.4 [10.2 to 24.4] | 14.9 [8.9 to 22.8] | 16.2 [10.1 to 24.2]
  Nausea: Moderate | 16.7 [10.3 to 24.8] | 8.7 [4.2 to 15.4] | 8.6 [4.2 to 15.3] | 4.4 [1.4 to 9.9] | 6.0 [2.4 to 11.9]
  Nausea: Severe | 0.9 [0.0 to 4.8] | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1]
  Muscle pain: Mild | 14.9 [8.9 to 22.8] | 28.7 [20.6 to 37.9] | 21.6 [14.5 to 30.1] | 21.9 [14.7 to 30.6] | 6.8 [3.0 to 13.0]
  Muscle pain: Moderate | 11.4 [6.2 to 18.7] | 14.8 [8.9 to 22.6] | 12.1 [6.8 to 19.4] | 14.0 [8.2 to 21.8] | 5.1 [1.9 to 10.8]
  Muscle pain: Severe | 0.9 [0.0 to 4.8] | 0.9 [0.0 to 4.7] | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1]
  Joint pain: Mild | 4.4 [1.4 to 9.9] | 7.8 [3.6 to 14.3] | 11.2 [6.1 to 18.4] | 7.0 [3.1 to 13.4] | 5.1 [1.9 to 10.8]
  Joint pain: Moderate | 9.6 [4.9 to 16.6] | 3.5 [1.0 to 8.7] | 9.5 [4.8 to 16.3] | 3.5 [1.0 to 8.7] | 4.3 [1.4 to 9.7]
  Joint pain: Severe | 0.9 [0.0 to 4.8] | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1]
  Vomiting: Mild | 11.4 [6.2 to 18.7] | 7.8 [3.6 to 14.3] | 5.2 [1.9 to 10.9] | 4.4 [1.4 to 9.9] | 6.0 [2.4 to 11.9]
  Vomiting: Moderate | 5.3 [2.0 to 11.1] | 5.2 [1.9 to 11.0] | 1.7 [0.2 to 6.1] | 0.0 [0.0 to 3.2] | 1.7 [0.2 to 6.0]
  Vomiting: Severe | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1] | 0.0 [0.0 to 3.2] | 0.0 [0.0 to 3.1]
  Diarrhea: Mild | 9.6 [4.9 to 16.6] | 10.4 [5.5 to 17.5] | 9.5 [4.8 to 16.3] | 7.0 [3.1 to 13.4] | 12.0 [6.7 to 19.3]
  Diarrhea: Moderate | 3.5 [1.0 to 8.7] | 0.0 [0.0 to 3.2] | 1.7 [0.2 to 6.1] | 3.5 [1.0 to 8.7] | 1.7 [0.2 to 6.0]
  Diarrhea: Severe | 0.0 [0.0 to 3.2] | 0.9 [0.0 to 4.7] | 0.0 [0.0 to 3.1] | 0.9 [0.0 to 4.8] | 0.0 [0.0 to 3.1]

3. Primary Outcome: Percentage of Maternal Participants With Adverse Events (AEs) Within 1 Month After Vaccination
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AEs included both serious and non-serious adverse events. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect.
Time Frame: Within 1 month after vaccination
Population: Maternal safety population included all randomized maternal participants who received investigational product and were analyzed according to the investigational product they received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Maternal Participants: RSVpreF 120 mcg | Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide | Maternal Participants: RSVpreF 240 mcg | Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide | Maternal Participants: Placebo
Number analyzed (Participants) | 115 | 117 | 116 | 114 | 117
Percentage of participants | 22.6 [15.3 to 31.3] | 23.9 [16.5 to 32.7] | 30.2 [22.0 to 39.4] | 22.8 [15.5 to 31.6] | 24.8 [17.3 to 33.6]

4. Primary Outcome: Percentage of Maternal Participants With Serious Adverse Events (SAEs), Medically Attended Adverse Events (MAEs) and Obstetric Complications
Description: MAE was defined as a non-serious AE that results in an evaluation at a medical facility. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect. Obstetric complications were determined as per the study clinician's judgement.
Time Frame: From day of vaccination (Day 1) up to 12 months post-delivery
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Maternal Participants: RSVpreF 120 mcg | Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide | Maternal Participants: RSVpreF 240 mcg | Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide | Maternal Participants: Placebo
Number analyzed (Participants) | 115 | 117 | 116 | 114 | 117
Percentage of participants
  SAE | 6.1 [2.5 to 12.1] | 12.8 [7.4 to 20.3] | 12.9 [7.4 to 20.4] | 16.7 [10.3 to 24.8] | 12.0 [6.7 to 19.3]
  MAE | 20.0 [13.1 to 28.5] | 18.8 [12.2 to 27.1] | 15.5 [9.5 to 23.4] | 21.1 [14.0 to 29.7] | 17.1 [10.8 to 25.2]
  Obstetric complications | 23.5 [16.1 to 32.3] | 28.2 [20.3 to 37.3] | 30.2 [22.0 to 39.4] | 33.3 [24.8 to 42.8] | 32.5 [24.1 to 41.8]

5. Primary Outcome: Percentage of Infant Participants With Specific Birth Complications
Description: Specific birth complications included clavicle fracture, torticollis, cephalhematoma, premature baby, acute respiratory failure, meconium aspiration syndrome, neonatal pneumothorax, neonatal respiratory depression, neonatal respiratory distress, neonatal respiratory distress syndrome, neonatal respiratory failure, pneumothorax, respiratory distress, transient tachypnea of the newborn and subgaleal hemorrhage. Percentage of participants with any specific birth complications were reported in this outcome measure.
Time Frame: At birth
Population: Infant safety population included all infant participants who were born to vaccinated maternal participants and were analyzed according to the investigational product their mothers received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infant Participants: RSVpreF 120 mcg | Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide | Infant Participants: RSVpreF 240 mcg | Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide | Infant Participants: Placebo
Number analyzed (Participants) | 114 | 117 | 113 | 112 | 116
Percentage of participants | 7.9 [3.7 to 14.5] | 10.3 [5.4 to 17.2] | 8.8 [4.3 to 15.7] | 8.0 [3.7 to 14.7] | 9.5 [4.8 to 16.3]

6. Primary Outcome: Percentage of Infant Participants With Any AE Within 1 Month of Age
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AEs included both serious and non-serious adverse events. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect.
Time Frame: Within 1 month after birth
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infant Participants: RSVpreF 120 mcg | Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide | Infant Participants: RSVpreF 240 mcg | Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide | Infant Participants: Placebo
Number analyzed (Participants) | 114 | 117 | 113 | 112 | 116
Percentage of participants | 50.9 [41.3 to 60.4] | 47.0 [37.7 to 56.5] | 46.9 [37.5 to 56.5] | 49.1 [39.5 to 58.7] | 50.9 [41.4 to 60.3]

7. Primary Outcome: Percentage of Infant Participants With MAEs and SAEs Within 12 Months of Age
Description: MAE was defined as a non-serious AE that results in an evaluation at a medical facility. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect.
Time Frame: Within 12 months after birth
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infant Participants: RSVpreF 120 mcg | Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide | Infant Participants: RSVpreF 240 mcg | Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide | Infant Participants: Placebo
Number analyzed (Participants) | 114 | 117 | 113 | 112 | 116
Percentage of participants
  MAE | 22.8 [15.5 to 31.6] | 29.9 [21.8 to 39.1] | 30.1 [21.8 to 39.4] | 38.4 [29.4 to 48.1] | 31.9 [23.6 to 41.2]
  SAE | 36.0 [27.2 to 45.5] | 33.3 [24.9 to 42.6] | 31.0 [22.6 to 40.4] | 39.3 [30.2 to 49.0] | 32.8 [24.3 to 42.1]

8. Primary Outcome: Percentage of Infant Participants With AEs of Special Interest of at Least Moderate Severity Within 12 Months of Age: Congenital Anomalies and Developmental Delay
Description: AEs of special interest for infant participants included congenital anomalies and developmental delays. Congenital anomalies were defined as structural or functional anomalies that occurred during intrauterine life and could be identified prenatally, at birth or later in life. Severity was assessed based on the study investigator's judgement and graded as grade 1= mild (does not interfere with participant's usual function); grade 2= moderate (interferes to some extent with participant's usual function); grade 3= severe (interferes significantly with participant's usual function) and grade 4= life-threatening (life-threatening consequences; urgent intervention indicated). Percentage of infant participants with AEs of special interest of at least moderate severity were presented.
Time Frame: Within 12 months after birth
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Infant Participants: RSVpreF 120 mcg | Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide | Infant Participants: RSVpreF 240 mcg | Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide | Infant Participants: Placebo
Number analyzed (Participants) | 114 | 117 | 113 | 112 | 116
Percentage of participants
  Congenital Anomalies | 9.6 [4.9 to 16.6] | 4.3 [1.4 to 9.7] | 1.8 [0.2 to 6.2] | 1.8 [0.2 to 6.3] | 6.0 [2.5 to 12.0]
  Developmental Delay | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

9. Secondary Outcome: Geometric Mean Titer (GMT) of Respiratory Syncytial Virus Subgroup A (RSV A) and Subgroup B (RSV B) Neutralizing Antibodies in Maternal Participants
Description: GMT of the 50% RSV A and RSV B neutralizing antibody were calculated by exponentiating the mean logarithm of the titers and the corresponding 95% confidence interval (CI) was based on the Student t distribution. Geometric mean ratios (GMRs) of the RSV vaccine group to the placebo group for the RSV A and RSV B neutralizing antibody titers at each time point was calculated and reported in statistical analysis.
Time Frame: Before vaccination, 2 weeks and 1 month after vaccination and at delivery
Population: Maternal evaluable immunogenicity population: eligible maternal participants who received randomized vaccine, had blood collection within protocol-specified time points, had at least 1 valid and determinate assay result after vaccination and had no other major protocol deviations. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies participants evaluable for this outcome measure at specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Maternal Participants: RSVpreF 120 mcg | Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide | Maternal Participants: RSVpreF 240 mcg | Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide | Maternal Participants: Placebo
Number analyzed (Participants) | 111 | 112 | 112 | 110 | 115
Titer
  A 50%: Before vaccination: number analyzed (Participants) | 111 | 112 | 112 | 110 | 114
  A 50%: Before vaccination | 1574 [1369.2 to 1808.7] | 1577 [1343.2 to 1850.9] | 1432 [1221.3 to 1678.2] | 1521 [1318.6 to 1754.4] | 1450 [1263.5 to 1663.3]
  A 50%: 2 Weeks after vaccination: number analyzed (Participants) | 102 | 100 | 99 | 101 | 104
  A 50%: 2 Weeks after vaccination | 31871 [27687.5 to 36685.8] | 31644 [25759.8 to 38873.3] | 33532 [28298.3 to 39733.8] | 39874 [33992.0 to 46773.6] | 1597 [1357.6 to 1879.4]
  A 50%: 1 Month after vaccination: number analyzed (Participants) | 102 | 98 | 97 | 96 | 97
  A 50%: 1 Month after vaccination | 24149 [19744.0 to 29537.1] | 31007 [26875.8 to 35773.7] | 23692 [19234.9 to 29182.2] | 28106 [24409.9 to 32362.2] | 1549 [1294.9 to 1853.7]
  A 50%: At delivery: number analyzed (Participants) | 107 | 109 | 103 | 103 | 111
  A 50%: At delivery | 12914 [10781.2 to 15469.2] | 17259 [14982.9 to 19881.3] | 12231 [9925.5 to 15071.8] | 15814 [13512.2 to 18507.5] | 1150 [957.4 to 1380.3]
  B 50%: Before vaccination | 1756 [1513.0 to 2038.3] | 1756 [1475.2 to 2090.8] | 1647 [1387.5 to 1955.6] | 1792 [1510.8 to 2125.2] | 1652 [1419.8 to 1923.2]
  B 50%: 2 Weeks after vaccination: number analyzed (Participants) | 102 | 100 | 99 | 101 | 104
  B 50%: 2 Weeks after vaccination | 39152 [31938.0 to 47996.6] | 36382 [28841.0 to 45893.9] | 43030 [35419.6 to 52275.2] | 55967 [46848.7 to 66861.1] | 1615 [1354.4 to 1926.1]
  B 50%: 1 Month after vaccination: number analyzed (Participants) | 102 | 98 | 97 | 96 | 97
  B 50%: 1 Month after vaccination | 34397 [28139.5 to 42046.9] | 37931 [31958.7 to 45019.8] | 30339 [23978.7 to 38387.3] | 39055 [32898.8 to 46363.2] | 1686 [1415.4 to 2007.3]
  B 50%: At delivery: number analyzed (Participants) | 107 | 109 | 103 | 103 | 111
  B 50%: At delivery | 16157 [12864.8 to 20291.4] | 19952 [16221.3 to 24540.1] | 16011 [12916.4 to 19847.7] | 19130 [15276.7 to 23955.2] | 1184 [977.1 to 1435.7]
Statistical Analysis 1: Comparison: Maternal Participants: RSVpreF 120 mcg vs Maternal Participants: Placebo; A 50%: Before vaccination; Test type: Other; Geometric Mean Ratio = 1.1, 95% CI 2-sided [0.9 to 1.3] — GMRs and 2-sided CIs were calculated by exponentiating the mean differences in the logarithms of the titers (RSV group - placebo group) and the corresponding CIs (CIs based on the Student t distribution)
Statistical Analysis 2: Comparison: Maternal Participants: RSVpreF 120 mcg vs Maternal Participants: Placebo; A 50%: 2 Weeks after vaccination; Test type: Other; Geometric Mean Ratio = 20.0, 95% CI 2-sided [16.1 to 24.7] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Maternal Participants: RSVpreF 120 mcg vs Maternal Participants: Placebo; A 50%: 1 Month after vaccination; Test type: Other; Geometric Mean Ratio = 15.6, 95% CI 2-sided [11.9 to 20.4] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Maternal Participants: RSVpreF 120 mcg vs Maternal Participants: Placebo; A 50%: At delivery; Test type: Other; Geometric Mean Ratio = 11.2, 95% CI 2-sided [8.7 to 14.5] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Maternal Participants: RSVpreF 120 mcg vs Maternal Participants: Placebo; B 50%: Before vaccination; Test type: Other; Geometric Mean Ratio = 1.1, 95% CI 2-sided [0.9 to 1.3] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Maternal Participants: RSVpreF 120 mcg vs Maternal Participants: Placebo; B 50%: 2 Weeks after vaccination; Test type: Other; Geometric Mean Ratio = 24.2, 95% CI 2-sided [18.5 to 31.7] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 7: Comparison: Maternal Participants: RSVpreF 120 mcg vs Maternal Participants: Placebo; B 50%: 1 Month after vaccination; Test type: Other; Geometric Mean Ratio = 20.4, 95% CI 2-sided [15.7 to 26.6] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 8: Comparison: Maternal Participants: RSVpreF 120 mcg vs Maternal Participants: Placebo; B 50%: At delivery; Test type: Other; Geometric Mean Ratio = 13.6, 95% CI 2-sided [10.1 to 18.4] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 9: Comparison: Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide vs Maternal Participants: Placebo; A 50%: Before vaccination; Test type: Other; Geometric Mean Ratio = 1.1, 95% CI 2-sided [0.9 to 1.3] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 10: Comparison: Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide vs Maternal Participants: Placebo; A 50%: 2 Weeks after vaccination; Test type: Other; Geometric Mean Ratio = 19.8, 95% CI 2-sided [15.3 to 25.7] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 11: Comparison: Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide vs Maternal Participants: Placebo; A 50%: 1 Month after vaccination; Test type: Other; Geometric Mean Ratio = 20.0, 95% CI 2-sided [15.9 to 25.1] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 12: Comparison: Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide vs Maternal Participants: Placebo; A 50%: At delivery; Test type: Other; Geometric Mean Ratio = 15.0, 95% CI 2-sided [11.9 to 18.9] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 13: Comparison: Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide vs Maternal Participants: Placebo; B 50%: Before vaccination; Test type: Other; Geometric Mean Ratio = 1.1, 95% CI 2-sided [0.8 to 1.3] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 14: Comparison: Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide vs Maternal Participants: Placebo; B 50%: 2 Weeks after vaccination; Test type: Other; Geometric Mean Ratio = 22.5, 95% CI 2-sided [16.9 to 30.1] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 15: Comparison: Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide vs Maternal Participants: Placebo; B 50%: 1 Month after vaccination; Test type: Other; Geometric Mean Ratio = 22.5, 95% CI 2-sided [17.6 to 28.7] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 16: Comparison: Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide vs Maternal Participants: Placebo; B 50%: At delivery; Test type: Other; Geometric Mean Ratio = 16.8, 95% CI 2-sided [12.7 to 22.3] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 17: Comparison: Maternal Participants: RSVpreF 240 mcg vs Maternal Participants: Placebo; A 50%: Before vaccination; Test type: Other; Geometric Mean Ratio = 1.0, 95% CI 2-sided [0.8 to 1.2] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 18: Comparison: Maternal Participants: RSVpreF 240 mcg vs Maternal Participants: Placebo; A 50%: 2 Weeks after vaccination; Test type: Other; Geometric Mean Ratio = 21.0, 95% CI 2-sided [16.6 to 26.5] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 19: Comparison: Maternal Participants: RSVpreF 240 mcg vs Maternal Participants: Placebo; A 50%: 1 Month after vaccination; Test type: Other; Geometric Mean Ratio = 15.3, 95% CI 2-sided [11.6 to 20.1] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 20: Comparison: Maternal Participants: RSVpreF 240 mcg vs Maternal Participants: Placebo; A 50%: At delivery; Test type: Other; Geometric Mean Ratio = 10.6, 95% CI 2-sided [8.1 to 14.0] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 21: Comparison: Maternal Participants: RSVpreF 240 mcg vs Maternal Participants: Placebo; B 50%: Before vaccination; Test type: Other; Geometric Mean Ratio = 1.0, 95% CI 2-sided [0.8 to 1.3] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 22: Comparison: Maternal Participants: RSVpreF 240 mcg vs Maternal Participants: Placebo; B 50%: 2 Weeks after vaccination; Test type: Other; Geometric Mean Ratio = 26.6, 95% CI 2-sided [20.5 to 34.6] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 23: Comparison: Maternal Participants: RSVpreF 240 mcg vs Maternal Participants: Placebo; B 50%: 1 Month after vaccination; Test type: Other; Geometric Mean Ratio = 18.0, 95% CI 2-sided [13.5 to 24.1] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 24: Comparison: Maternal Participants: RSVpreF 240 mcg vs Maternal Participants: Placebo; B 50%: At delivery; Test type: Other; Geometric Mean Ratio = 13.5, 95% CI 2-sided [10.1 to 18.0] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 25: Comparison: Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide vs Maternal Participants: Placebo; A 50%: Before vaccination; Test type: Other; Geometric Mean Ratio = 1.0, 95% CI 2-sided [0.9 to 1.3] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 26: Comparison: Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide vs Maternal Participants: Placebo; A 50%: 2 Weeks after vaccination; Test type: Other; Geometric Mean Ratio = 25.0, 95% CI 2-sided [19.9 to 31.3] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 27: Comparison: Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide vs Maternal Participants: Placebo; A 50%: 1 Month after vaccination; Test type: Other; Geometric Mean Ratio = 18.1, 95% CI 2-sided [14.5 to 22.8] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 28: Comparison: Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide vs Maternal Participants: Placebo; A 50%: At delivery; Test type: Other; Geometric Mean Ratio = 13.8, 95% CI 2-sided [10.8 to 17.5] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 29: Comparison: Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide vs Maternal Participants: Placebo; B 50%: Before vaccination; Test type: Other; Geometric Mean Ratio = 1.1, 95% CI 2-sided [0.9 to 1.4] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 30: Comparison: Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide vs Maternal Participants: Placebo; B 50%: 2 Weeks after vaccination; Test type: Other; Geometric Mean Ratio = 34.7, 95% CI 2-sided [27.0 to 44.4] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 31: Comparison: Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide vs Maternal Participants: Placebo; B 50%: 1 Month after vaccination; Test type: Other; Geometric Mean Ratio = 23.2, 95% CI 2-sided [18.2 to 29.6] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 32: Comparison: Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide vs Maternal Participants: Placebo; B 50%: At delivery; Test type: Other; Geometric Mean Ratio = 16.2, 95% CI 2-sided [12.0 to 21.7] — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Geometric Mean Fold Rise (GMFR) for Respiratory Syncytial Virus Subgroup A (RSV A) and Subgroup B (RSV B) Neutralizing Antibody Titers in Maternal Participants
Description: GMFRs for RSV A and RSV B neutralizing antibody titers from before vaccination to each available time point after vaccination were calculated by exponentiating the mean logarithm of the fold rises. Corresponding 95% CI was based on the Student t distribution. Data for this outcome measure was planned to be analyzed for maternal participants only.
Time Frame: 2 weeks and 1 month after vaccination, at delivery
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Maternal Participants: RSVpreF 120 mcg | Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide | Maternal Participants: RSVpreF 240 mcg | Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide | Maternal Participants: Placebo
Number analyzed (Participants) | 106 | 108 | 103 | 103 | 111
Fold rise
  A 50%: 2 Weeks after vaccination: number analyzed (Participants) | 102 | 99 | 99 | 101 | 103
  A 50%: 2 Weeks after vaccination | 19.8 [16.35 to 24.04] | 20.4 [16.12 to 25.77] | 23.3 [19.27 to 28.10] | 25.3 [20.97 to 30.52] | 1.1 [0.95 to 1.28]
  A 50%: 1 Month after vaccination: number analyzed (Participants) | 102 | 97 | 97 | 96 | 96
  A 50%: 1 Month after vaccination | 14.9 [11.89 to 18.65] | 19.6 [16.21 to 23.61] | 15.9 [12.85 to 19.80] | 17.8 [14.99 to 21.04] | 1.0 [0.94 to 1.18]
  A 50%: At delivery: number analyzed (Participants) | 106 | 108 | 103 | 103 | 110
  A 50%: At delivery | 8.3 [6.85 to 10.05] | 10.9 [9.33 to 12.78] | 8.6 [6.81 to 10.74] | 10.6 [8.91 to 12.56] | 0.8 [0.67 to 0.95]
  B 50%: 2 Weeks after vaccination: number analyzed (Participants) | 102 | 99 | 99 | 101 | 104
  B 50%: 2 Weeks after vaccination | 21.8 [17.24 to 27.47] | 21.0 [16.69 to 26.35] | 26.4 [21.36 to 32.51] | 30.4 [24.35 to 37.83] | 1.0 [0.84 to 1.16]
  B 50%: 1 Month after vaccination: number analyzed (Participants) | 102 | 97 | 97 | 96 | 97
  B 50%: 1 Month after vaccination | 19.2 [15.43 to 23.84] | 22.0 [18.30 to 26.41] | 17.7 [13.94 to 22.51] | 20.9 [17.42 to 25.12] | 1.0 [0.90 to 1.17]
  B 50%: At delivery | 9.2 [7.19 to 11.74] | 11.2 [9.20 to 13.74] | 9.5 [7.80 to 11.48] | 10.7 [8.49 to 13.49] | 0.7 [0.61 to 0.87]

11. Secondary Outcome: Geometric Mean Titer (GMT) of Respiratory Syncytial Virus Subgroup A (RSV A) and Subgroup B (RSV B) Neutralizing Antibodies in Infant Participants
Description: GMT of the 50% RSV A and RSV B neutralizing antibody were calculated by exponentiating the mean logarithm of the titers and the corresponding 95% CI was based on the Student t distribution. GMRs of the RSV vaccine group to the placebo group for the RSV A and RSV B neutralizing antibody titers at each time point was calculated and reported in statistical analysis.
Time Frame: At birth and at 1, 2, 4, 6 months after birth
Population: Infant evaluable immunogenicity population: eligible infant participants born to maternal participants who received randomized vaccine and had no protocol deviation before delivery, had blood collection within protocol-specified time point at birth, had at least 1 valid, determinate assay result at birth and had no other major protocol deviations. Here, 'Number Analyzed' signifies participants evaluable for this outcome measure at specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Infant Participants: RSVpreF 120 mcg | Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide | Infant Participants: RSVpreF 240 mcg | Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide | Infant Participants: Placebo
Number analyzed (Participants) | 100 | 109 | 103 | 104 | 106
Titer
  A 50%: At birth: number analyzed (Participants) | 100 | 108 | 103 | 103 | 106
  A 50%: At birth | 22904 [18636.8 to 28147.5] | 23281 [19155.8 to 28294.3] | 20530 [17271.7 to 24403.0] | 24290 [19858.5 to 29710.2] | 2150 [1776.7 to 2602.6]
  A 50%: 1 Month after birth: number analyzed (Participants) | 37 | 37 | 33 | 41 | 30
  A 50%: 1 Month after birth | 13532 [8775.4 to 20865.4] | 14667 [10428.4 to 20627.6] | 12685 [9161.6 to 17563.9] | 15383 [12253.4 to 19311.4] | 1514 [1200.9 to 1908.0]
  A 50%: 2 Months after birth: number analyzed (Participants) | 27 | 35 | 37 | 35 | 40
  A 50%: 2 Months after birth | 11127 [8424.3 to 14695.8] | 7455 [5517.1 to 10073.8] | 6943 [4890.5 to 9858.0] | 10552 [8019.3 to 13884.7] | 702 [529.5 to 930.8]
  A 50%: 4 Months after birth: number analyzed (Participants) | 35 | 30 | 34 | 31 | 36
  A 50%: 4 Months after birth | 2673 [1904.5 to 3753.0] | 3919 [2905.9 to 5285.8] | 2148 [1681.5 to 2743.3] | 2936 [2217.6 to 3887.3] | 478 [336.3 to 680.2]
  A 50%: 6 Months after birth: number analyzed (Participants) | 35 | 39 | 40 | 29 | 39
  A 50%: 6 Months after birth | 1529 [1164.8 to 2008.3] | 1124 [790.0 to 1600.4] | 930 [643.0 to 1344.2] | 1048 [747.6 to 1468.5] | 233 [176.2 to 307.0]
  B 50%: At birth | 30195 [24308.9 to 37506.3] | 28437 [22968.2 to 35207.9] | 25112 [20172.4 to 31262.1] | 32967 [27494.5 to 39529.5] | 2029 [1669.5 to 2466.2]
  B 50%: 1 Month after birth: number analyzed (Participants) | 37 | 38 | 33 | 41 | 30
  B 50%: 1 Month after birth | 17418 [11133.3 to 27251.5] | 18708 [12994.4 to 26934.9] | 17911 [12397.2 to 25876.7] | 20353 [15477.7 to 26762.8] | 1586 [1181.0 to 2129.1]
  B 50%: 2 Months after birth: number analyzed (Participants) | 27 | 35 | 37 | 35 | 40
  B 50%: 2 Months after birth | 13411 [10016.5 to 17955.2] | 8341 [5847.7 to 11898.6] | 7251 [5387.9 to 9757.8] | 12359 [9060.4 to 16857.4] | 700 [542.3 to 903.6]
  B 50%: 4 Months after birth: number analyzed (Participants) | 35 | 30 | 35 | 31 | 36
  B 50%: 4 Months after birth | 3168 [2261.8 to 4436.5] | 4075 [2952.0 to 5624.6] | 2621 [2029.1 to 3385.5] | 4135 [3093.4 to 5526.2] | 458 [313.6 to 668.3]
  B 50%: 6 Months after birth: number analyzed (Participants) | 35 | 39 | 40 | 29 | 40
  B 50%: 6 Months after birth | 1609 [1094.5 to 2364.3] | 1195 [805.8 to 1772.0] | 956 [656.8 to 1392.7] | 1381 [966.6 to 1972.0] | 221 [162.9 to 300.9]
Statistical Analysis 1: Comparison: Infant Participants: RSVpreF 120 mcg vs Infant Participants: Placebo; A 50%: At birth; Test type: Other; Geometric Mean Ratio = 10.7, 95% CI 2-sided [8.1 to 14.1] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Infant Participants: RSVpreF 120 mcg vs Infant Participants: Placebo; A 50%: 1 Month after birth; Test type: Other; Geometric Mean Ratio = 8.9, 95% CI 2-sided [5.5 to 14.5] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Infant Participants: RSVpreF 120 mcg vs Infant Participants: Placebo; A 50%: 2 Months after birth; Test type: Other; Geometric Mean Ratio = 15.8, 95% CI 2-sided [10.7 to 23.4] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Infant Participants: RSVpreF 120 mcg vs Infant Participants: Placebo; A 50%: 4 Months after birth; Test type: Other; Geometric Mean Ratio = 5.6, 95% CI 2-sided [3.5 to 9.0] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 5: Comparison: Infant Participants: RSVpreF 120 mcg vs Infant Participants: Placebo; A 50%: 6 Months after birth; Test type: Other; Geometric Mean Ratio = 6.6, 95% CI 2-sided [4.5 to 9.6] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 6: Comparison: Infant Participants: RSVpreF 120 mcg vs Infant Participants: Placebo; B 50%: At birth; Test type: Other; Geometric Mean Ratio = 14.9, 95% CI 2-sided [11.1 to 19.9] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 7: Comparison: Infant Participants: RSVpreF 120 mcg vs Infant Participants: Placebo; B 50%: 1 Month after birth; Test type: Other; Geometric Mean Ratio = 11.0, 95% CI 2-sided [6.5 to 18.6] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 8: Comparison: Infant Participants: RSVpreF 120 mcg vs Infant Participants: Placebo; B 50%: 2 Months after birth; Test type: Other; Geometric Mean Ratio = 19.2, 95% CI 2-sided [13.1 to 28.0] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 9: Comparison: Infant Participants: RSVpreF 120 mcg vs Infant Participants: Placebo; B 50%: 4 Months after birth; Test type: Other; Geometric Mean Ratio = 6.9, 95% CI 2-sided [4.2 to 11.4] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 10: Comparison: Infant Participants: RSVpreF 120 mcg vs Infant Participants: Placebo; B 50%: 6 Months after birth; Test type: Other; Geometric Mean Ratio = 7.3, 95% CI 2-sided [4.5 to 11.8] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 11: Comparison: Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; A 50%: At birth; Test type: Other; Geometric Mean Ratio = 10.8, 95% CI 2-sided [8.3 to 14.2] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 12: Comparison: Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; A 50%: 1 Month after birth; Test type: Other; Geometric Mean Ratio = 9.7, 95% CI 2-sided [6.5 to 14.5] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 13: Comparison: Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; A 50%: 2 Months after birth; Test type: Other; Geometric Mean Ratio = 10.6, 95% CI 2-sided [7.1 to 15.9] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 14: Comparison: Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; A 50%: 4 Months after birth; Test type: Other; Geometric Mean Ratio = 8.2, 95% CI 2-sided [5.2 to 12.9] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 15: Comparison: Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; A 50%: 6 Months after birth; Test type: Other; Geometric Mean Ratio = 4.8, 95% CI 2-sided [3.1 to 7.5] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 16: Comparison: Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; B 50%: At birth; Test type: Other; Geometric Mean Ratio = 14.0, 95% CI 2-sided [10.5 to 18.7] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 17: Comparison: Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; B 50%: 1 Month after birth; Test type: Other; Geometric Mean Ratio = 11.8, 95% CI 2-sided [7.4 to 18.7] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 18: Comparison: Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; B 50%: 2 Months after birth; Test type: Other; Geometric Mean Ratio = 11.9, 95% CI 2-sided [7.7 to 18.3] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 19: Comparison: Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; B 50%: 4 Months after birth; Test type: Other; Geometric Mean Ratio = 8.9, 95% CI 2-sided [5.5 to 14.5] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 20: Comparison: Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; B 50%: 6 Months after birth; Test type: Other; Geometric Mean Ratio = 5.4, 95% CI 2-sided [3.3 to 8.8] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 21: Comparison: Infant Participants: RSVpreF 240 mcg vs Infant Participants: Placebo; A 50%: At birth; Test type: Other; Geometric Mean Ratio = 9.5, 95% CI 2-sided [7.4 to 12.3] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 22: Comparison: Infant Participants: RSVpreF 240 mcg vs Infant Participants: Placebo; A 50%: 1 Month after birth; Test type: Other; Geometric Mean Ratio = 8.4, 95% CI 2-sided [5.7 to 12.4] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 23: Comparison: Infant Participants: RSVpreF 240 mcg vs Infant Participants: Placebo; A 50%: 2 Months after birth; Test type: Other; Geometric Mean Ratio = 9.9, 95% CI 2-sided [6.4 to 15.4] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 24: Comparison: Infant Participants: RSVpreF 240 mcg vs Infant Participants: Placebo; A 50%: 4 Months after birth; Test type: Other; Geometric Mean Ratio = 4.5, 95% CI 2-sided [2.9 to 6.8] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 25: Comparison: Infant Participants: RSVpreF 240 mcg vs Infant Participants: Placebo; A 50%: 6 Months after birth; Test type: Other; Geometric Mean Ratio = 4.0, 95% CI 2-sided [2.5 to 6.3] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 26: Comparison: Infant Participants: RSVpreF 240 mcg vs Infant Participants: Placebo; B 50%: At birth; Test type: Other; Geometric Mean Ratio = 12.4, 95% CI 2-sided [9.2 to 16.6] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 27: Comparison: Infant Participants: RSVpreF 240 mcg vs Infant Participants: Placebo; B 50%: 1 Month after birth; Test type: Other; Geometric Mean Ratio = 11.3, 95% CI 2-sided [7.1 to 17.9] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 28: Comparison: Infant Participants: RSVpreF 240 mcg vs Infant Participants: Placebo; B 50%: 2 Months after birth; Test type: Other; Geometric Mean Ratio = 10.4, 95% CI 2-sided [7.0 to 15.2] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 29: Comparison: Infant Participants: RSVpreF 240 mcg vs Infant Participants: Placebo; B 50%: 4 Months after birth; Test type: Other; Geometric Mean Ratio = 5.7, 95% CI 2-sided [3.7 to 9.0] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 30: Comparison: Infant Participants: RSVpreF 240 mcg vs Infant Participants: Placebo; B 50%: 6 Months after birth; Test type: Other; Geometric Mean Ratio = 4.3, 95% CI 2-sided [2.7 to 7.0] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 31: Comparison: Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; A 50%: At birth; Test type: Other; Geometric Mean Ratio = 11.3, 95% CI 2-sided [8.6 to 14.9] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 32: Comparison: Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; A 50%: 1 Month after birth; Test type: Other; Geometric Mean Ratio = 10.2, 95% CI 2-sided [7.4 to 14.0] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 33: Comparison: Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; A 50%: 2 Months after birth; Test type: Other; Geometric Mean Ratio = 15.0, 95% CI 2-sided [10.2 to 22.1] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 34: Comparison: Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; A 50%: 4 Months after birth; Test type: Other; Geometric Mean Ratio = 6.1, 95% CI 2-sided [3.9 to 9.6] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 35: Comparison: Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; A 50%: 6 Months after birth; Test type: Other; Geometric Mean Ratio = 4.5, 95% CI 2-sided [2.9 to 6.9] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 36: Comparison: Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; B 50%: At birth; Test type: Other; Geometric Mean Ratio = 16.2, 95% CI 2-sided [12.5 to 21.2] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 37: Comparison: Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; B 50%: 1 Month after birth; Test type: Other; Geometric Mean Ratio = 12.8, 95% CI 2-sided [8.6 to 19.1] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 38: Comparison: Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; B 50%: 2 Months after birth; Test type: Other; Geometric Mean Ratio = 17.7, 95% CI 2-sided [11.9 to 26.2] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 39: Comparison: Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; B 50%: 4 Months after birth; Test type: Other; Geometric Mean Ratio = 9.0, 95% CI 2-sided [5.7 to 14.4] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 40: Comparison: Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide vs Infant Participants: Placebo; B 50%: 6 Months after birth; Test type: Other; Geometric Mean Ratio = 6.2, 95% CI 2-sided [3.9 to 9.9] — [estimate comment as in outcome 9, analysis 1]

ADVERSE EVENTS:
Time Frame: Local reactions and systematic events (systematic assessment): within 7 days after vaccination. AEs and SAEs (non-systematic assessment): From day of vaccination (Day 1) up to 12 months post-delivery for maternal participants and from birth up to 12 months after birth for infant participants
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Maternal safety population was evaluated for maternal participants and Infant safety population for infant participants.
Arm/Group | Maternal Participants: RSVpreF 120 mcg | Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide | Maternal Participants: RSVpreF 240 mcg | Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide | Maternal Participants: Placebo | Infant Participants: RSVpreF 120 mcg | Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide | Infant Participants: RSVpreF 240 mcg | Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide | Infant Participants: Placebo
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/117 | 0/116 | 0/114 | 0/117 | 0/114 | 0/117 | 0/113 | 0/112 | 0/116
Serious Adverse Events (participants affected / at risk) | 7/115 | 15/117 | 15/116 | 19/114 | 14/117 | 41/114 | 39/117 | 35/113 | 44/112 | 38/116
Other Adverse Events (participants affected / at risk) | 87/115 | 108/117 | 96/116 | 103/114 | 89/117 | 66/114 | 59/117 | 67/113 | 66/112 | 71/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Maternal Participants: RSVpreF 120 mcg (N=115) | Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide (N=117) | Maternal Participants: RSVpreF 240 mcg (N=116) | Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide (N=114) | Maternal Participants: Placebo (N=117) | Infant Participants: RSVpreF 120 mcg (N=114) | Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide (N=117) | Infant Participants: RSVpreF 240 mcg (N=113) | Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide (N=112) | Infant Participants: Placebo (N=116)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Baseline foetal heart rate variability disorder (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foetal heart rate deceleration abnormality (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nonreassuring foetal heart rate pattern (Cardiac disorders) | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia foetal (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Amniotic cavity infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anorectal cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Endometritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Endometritis decidual (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mastitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oophoritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Salpingitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uterine rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Foetal heart rate decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foetal heart rate indeterminate (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza virus test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
False labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 3 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical cord abnormality (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine tachysystole (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alpers disease (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 4 | 3 | 4
Aplasia cutis congenita (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1
Birth mark (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Chordee (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Chromosomal deletion (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cleft lip (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cleft palate (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Congenital coronary artery malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Congenital naevus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 6 | 9 | 3
Congenital skin dimples (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Congenital tracheomalacia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Congenital umbilical hernia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 6 | 1 | 3
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 1
Cystic fibrosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Double ureter (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal disorder congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoglobin D trait (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 2
Hypospadias (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0
Labial tie (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Laryngomalacia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Naevus flammeus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 4 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Penile torsion (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Penoscrotal fusion (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Polydactyly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spina bifida cystica (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Supernumerary nipple (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
XYY syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingival cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tongue cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 5 | 5 | 7 | 6
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 0
Adenovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Postoperative adhesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acoustic stimulation tests abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Cardiac murmur functional (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory syncytial virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Right ventricular systolic pressure (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Brain hypoxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clonic convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Encephalopathy neonatal (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Testicular retraction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cafe au lait spots (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subgaleal haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Neonatal aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neonatal pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neonatal respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Maternal Participants: RSVpreF 120 mcg (N=115) | Maternal Participants: RSVpreF 120 mcg With Aluminum Hydroxide (N=117) | Maternal Participants: RSVpreF 240 mcg (N=116) | Maternal Participants: RSVpreF 240 mcg With Aluminum Hydroxide (N=114) | Maternal Participants: Placebo (N=117) | Infant Participants: RSVpreF 120 mcg (N=114) | Infant Participants: RSVpreF 120 mcg With Aluminum Hydroxide (N=117) | Infant Participants: RSVpreF 240 mcg (N=113) | Infant Participants: RSVpreF 240 mcg With Aluminum Hydroxide (N=112) | Infant Participants: Placebo (N=116)
Anaemia (Blood and lymphatic system disorders) | 2 | 4 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nonreassuring foetal heart rate pattern (Cardiac disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 0 | 4 | 1 | 2 | 0 | 0
Diarrhoea (DIARRHOEA) (Gastrointestinal disorders) | 15 | 13 | 13 | 13 | 16 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3 | 1 | 1 | 0 | 3 | 4 | 6 | 7 | 9
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 4 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Nausea (NAUSEA) (Gastrointestinal disorders) | 37 | 31 | 29 | 22 | 26 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 1
Vomiting (VOMITING) (Gastrointestinal disorders) | 19 | 15 | 8 | 5 | 9 | 0 | 0 | 0 | 0 | 0
Fatigue (FATIGUE) (General disorders) | 55 | 55 | 53 | 58 | 55 | 0 | 0 | 0 | 0 | 0
Injection site erythema (REDNESS) (General disorders) | 5 | 5 | 7 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Injection site pain (PAIN AT INJECTION SITE) (General disorders) | 33 | 81 | 40 | 69 | 15 | 0 | 0 | 0 | 0 | 0
Injection site swelling (SWELLING) (General disorders) | 4 | 6 | 6 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0 | 5 | 5 | 5 | 4 | 3
Pyrexia (FEVER) (General disorders) | 4 | 6 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial disease carrier (Infections and infestations) | 2 | 4 | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 3 | 0 | 0 | 1 | 2
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 1 | 0
Mastitis (Infections and infestations) | 0 | 2 | 3 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 3 | 0 | 2 | 7 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 3 | 3 | 0 | 24 | 21 | 19 | 15 | 16
Urinary tract infection (Infections and infestations) | 3 | 3 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Perineal injury (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial test positive (Investigations) | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Streptococcus test positive (Investigations) | 5 | 5 | 2 | 5 | 4 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 17 | 14 | 24 | 12 | 11 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4 | 2 | 0 | 0 | 0 | 0 | 0
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 31 | 51 | 40 | 41 | 14 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Headache (HEADACHE) (Nervous system disorders) | 33 | 43 | 43 | 33 | 30 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 2 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 6 | 2 | 7 | 4 | 2 | 0 | 0 | 0 | 0 | 0
Shoulder dystocia (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Perinatal depression (Psychiatric disorders) | 5 | 2 | 2 | 4 | 2 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 0 | 7 | 7 | 4 | 6 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3 | 8 | 4 | 9 | 8 | 8
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0 | 1 | 5 | 0 | 3 | 6
Hypertension (Vascular disorders) | 3 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 4
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 4 | 3 | 3
Teething (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 6 | 2 | 10 | 4
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 12 | 7 | 8 | 6 | 5
Acne infantile (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 3 | 3 | 3
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 4 | 2 | 2
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Acquired plagiocephaly (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 5
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 2
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 7 | 3 | 1
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 10 | 10 | 8 | 10 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 2 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 6 | 3 | 3 | 2 | 4
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 4 | 2
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 3 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 5 | 3
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 4 | 6 | 9
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 5 | 3 | 6 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 3 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/93/NCT04032093/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT04032093/SAP_001.pdf